CLINICAL TRIAL: NCT04922385
Title: Cognitive Behavioural Therapy for Sexual Concerns During Perimenopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Sheryl Green, Clinical Psychologist, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBT-SC-Peri
Record Dates: First submitted 2021-06-06; First posted 2021-06-10 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Perimenopause; Sexual Concerns
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT (Experimental): Individual 4-week CBT protocol
  Interventions: Other: Cognitive Behavioural Therapy

INTERVENTIONS:
Other: Cognitive Behavioural Therapy — This study is an open waitlist control study. Eligible participants will be assigned to a treating clinician and will complete 4 weeks of treatment, followed by a post-treatment assessment (2 weeks later). If a treating clinician is not immediately available, participants will be placed on their waitlist for 4 weeks. They will then be assessed after 4 weeks and undergo the 4 week treatment, followed by the post-treatment assessment (2 weeks later).

SUMMARY:
Given the high rates and associated impairment of sexual concerns during the menopausal transition, and specifically during perimenopause, our team has developed a CBT protocol specifically designed to target these prevalent and distressing sexual concerns. The broad aim of the proposed study is to validate this new protocol in a clinic that provides empirically-supported assessment and intervention services for women with menopause-related symptoms. The primary objective of this study is to evaluate the efficacy of a four-week individual CBT protocol in improving sexual satisfaction and reducing distress during perimenopause. The secondary objective of this study is to evaluate the efficacy of this CBT protocol to improve sexual functioning (e.g., desire, arousal), relationship satisfaction, and body image. Exploratory analyses will examine the impact on this CBT protocol on vasomotor symptoms, depression, and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. 40-60 years of age;
2. peri-menopausal and have had a menstrual period within the previous twelve months as per the STRAW definition (Harlow et al., 2012);
3. cut-off score of 26 or lower on the Female Sexual Functioning Index, indicating sexual dysfunction (Wiegel et al., 2005);
4. medication stable (e.g., hormone therapy), with no changes in dosing for the previous three months (Green et al., 2019);
5. no psychological treatment to address sexual dysfunction and/or sexual concerns within the previous six months; and
6. speak, read, and write in English to comprehend testing procedures and written materials in treatment
7. living within Canada

Exclusion Criteria:

1. participants with psychotic disorders, or current substance and/or alcohol dependence; and
2. participants who are severely depressed/suicidal at time of the intake assessment.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Female Sexual Desire Questionnaire (FSDQ) | 6 weeks
  The FSDQ (Goldhammer & McCabe, 2011) is a 50-item self-report questionnaire assessing one's experience of and sexual desire for women across six domains: dyadic desire, solitary desire, resistance, positive relationship, sexual self-image, and concern. Total scores range from 50 to 300, with higher scores indicated increased sexual desire.
Female Sexual Distress Scale-Revised (FSDS-R) | 6 weeks
  The FSDS-R (DeRogatis et al., 2008) is a 13-item self-report questionnaire assessing various aspects of sexual distress, with a clinical cut-off score of 11 indicated sexual distress. Scores on the FSDS-R range from 0 to 48, with higher scores indicating greater sexual distress.
The Female Sexual Function Index (FSFI) | 6 weeks
  The FSFI (Rosen et al., 2000) is a six domain measure of female sexual functioning including sexual desire, subjective arousal, lubrication, orgasm, satisfaction, and pain. Scores on the FSFI range from 2-36, which higher scores indicating a greater level of sexual function.

SECONDARY OUTCOMES:
The Greene Climacteric Scale (GCS) | 6 weeks
  The GCS (Greene, 1998) is a self-report questionnaire measuring four menopause-related domains: vasomotor symptoms, depression and anxiety, physical complaints, and sexual concerns. Studies have shown women who score greater than 12 on the GCS are more likely to be menopausal.
The Hot Flash Related Daily Interference Scale (HFRDIS) | 6 weeks
  The HFRDIS (Carpenter, 2001) assesses the degree to which vasomotor symptoms interfere with daily life. Higher scores on the HFRDIS indicate higher interference due to hot flashes and thus, greater impact on quality of life.
The Beck Depression Inventory-II (BDI-II) | 6 weeks
  The BDI-II (Beck et al., 1996) is a self-report questionnaire and one of the most widely used tools for measuring depression. Total scores on the BDI-II range from 0-63, with higher scores indicating increased depressive symptom severity.
The Hamilton Anxiety Scale (HAM-A) | 6 weeks
  The HAM-A (Hamilton, 1959) is a clinician administered questionnaire developed to quantify the severity of anxiety symptomatology and is considered a gold-standard. Total scores on the HAM-A range from 0-56, with greater scores indicating increased anxiety severity.
The Couples Satisfaction Index (CSI) | 6 weeks
  The CSI (Funk & Rogge, 2007) is a 32-item scale designed to measure one's satisfaction in a relationship. Total scores on the CSI range from 0-81, with higher scores indicating greater couples satisfaction.
36-Item Short-Form Health Survey (SF-36) | 6 weeks
  The SF-36 (Ware & Sherbourne, 1992) is a 36-item self-administered questionnaire assessing one's perception of overall health and well-being. Higher scores on each domain indicate a more favourable health state in that area.
Dresden Body Image Questionnaire (DBIQ) | 6 weeks
  The DBIQ (Scheffers et al., 2017) is a 35-item self-report questionnaire assessing one's feelings of their physical appearance across five subscales: body acceptance, sexual fulfillment, physical contact, vitality, and self-aggrandizement. Higher score on the DBIQ indicate a more positive body image.
Cognitive Flexibility Inventory (CFI) | 6 weeks
  The CFI (Dennis & Vander Wal, 2010) is a 20-item self-report questionnaire that assesses three aspects of cognitive flexibility: tendency to perceive difficult situations as controllable, ability to perceive multiple alternative explanations for life occurrences and human behaviour, and ability to generate multiple alternative solutions to difficult situations. Higher scores are indicative of greater cognitive flexibility when encountering stressful situations.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl M Green, PhD, CPsych, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green SM, Furtado M, Shea AK, Ballantyne EC, Streiner DL, Frey BN, McCabe RE. Cognitive behavioural therapy for sexual concerns during menopause: evaluation of a four session protocol. J Sex Med. 2025 Jun 29;22(7):1184-1195. doi: 10.1093/jsxmed/qdaf085. PMID 40384525
- [Derived] Green SM, Furtado M. Cognitive Behavioral Therapy for Sexual Concerns During Perimenopause: A Four Session Study Protocol. Front Glob Womens Health. 2021 Oct 6;2:744748. doi: 10.3389/fgwh.2021.744748. eCollection 2021. PMID 34816248